CLINICAL TRIAL: NCT03743545
Title: ASSESSEMENT OF LOW SPEED DRILLING WITHOUT IRRIGATION VERSUS CONVENTIONEL DRILLING WITH IRRIGATION REGARDING HEAT GENERATION AND PERI-IMPLANT MARGINAL BONE LOSS
Brief Title: Assessment of Heat Generation From Low Speed Drilling Without Irrigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel Sattar Abdel Motagly, director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28601270201414
Record Dates: First submitted 2018-11-04; First posted 2018-11-16 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Implant Site Reaction
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: healthy posterior mandible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional drilling with irrigation (Active Comparator)
  Interventions: Other: low speed drilling without irrigation
- low speed without irrigation (Experimental)
  Interventions: Other: low speed drilling without irrigation

INTERVENTIONS:
Other: low speed drilling without irrigation — comparing between conventional implant placement drilling speed with irrigation and experimental arm (low speed without irrigation)

SUMMARY:
ASSESSMENT OF LOW SPEED DRILLING WITHOUT IRRIGATION VERSUS CONVENTIONAL DRILLING WITH IRRIGATION REGARDING HEAT GENERATION AND PERI-IMPLANT MARGINAL BONE LOSS

DETAILED DESCRIPTION:
Assessment of heat generation from conventional drilling speed for dental implant placement versus biological drilling (low speed without irrigation ) by thermocouples technology And measure the primary stability of dental implants placed by the two techniques by osstel device

ELIGIBILITY:
Inclusion Criteria: both sex no intraoral soft and hard tissue pathology no systemic condition that contraindicate implant placement adult patients with proper posterior mandibular ridge requires implant placement

Exclusion Criteria:

presence of pathological lesions heavy smokers more than 20 cigarettes per day patients with systemic disease that may affect normal healing Patients with no enough bone in posterior mandible for implant placement

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of heat generation from low speed hand piece drills drilling by thermocouple technology | 6 months
  Measurement of 3 different depths(mms). Data analyzed with a three-way analysis of variance by Newman-Keulsmultiple comparison procedure. The significance level was set to a p-value of 0.05.

SECONDARY OUTCOMES:
stability-osstell device to assess the primary stability of placed dental implant | 6 months
  Resonance frequency analysis (RFA) allows assess implant stability by measuring implant oscillation frequency on the bone